CLINICAL TRIAL: NCT01614613
Title: Clinical Evaluation of Bayer G3 / Tatsu System and BGMs From Other Companies
Brief Title: Comparison Evaluation of Blood Glucose Meter Systems in a Clinical Setting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ascensia Diabetes Care (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CTD-2010-009-02
Record Dates: First submitted 2012-05-13; First posted 2012-06-08 (Estimated); Results first posted 2013-09-09 (Estimated); Last update posted 2016-02-29 (Estimated); Status verified 2016-01

CONDITIONS: Diabetes
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Intended BGM Users (Experimental): Subjects were assigned to subgroups according to their initial glucose levels. SUBGROUP 1 goal: safely decrease subject glucose levels during the visit. SUBGROUP 2 goal: safely raise subject glucose levels. Also, blood samples were modified to obtain glucose concentrations across the needed glucose ranges while maintaining subject safety. Staff tested the blood samples using the 6 Blood Glucose Monitoring Systems. Bayer G3/Tatsu System;Accu-Chek® Aviva Nano Meter/Accu-Chek® Aviva Test Strips; Freestyle Lite® Meter and Test Strips with ZipwikTM tabs;OneTouch® Ultra®2 / OneTouch® Ultra® Blue Test Strips;One Touch® VerioTM Pro/One Touch® VerioTM Test Strips;Truetrack® Meter/Truetrack® Test Strips
  Interventions: Device: Bayer G3 / Tatsu System; Device: Accu-Chek® Aviva Nano Meter/Accu-Chek® Aviva Test Strips; Device: Freestyle Lite® Meter and Test Strips with ZipwikTM tabs; Device: OneTouch® Ultra®2 / OneTouch® Ultra® Blue Test Strips; Device: One Touch® VerioTM Pro/One Touch® VerioTM Test Strips; Device: Truetrack® Meter/Truetrack® Test Strips

INTERVENTIONS:
Device: Bayer G3 / Tatsu System — Study staff performed Blood Glucose (BG) tests with capillary fingerstick blood collected from subjects with diabetes. All meter BG results were compared with plasma results obtained with a reference laboratory glucose method (YSI Glucose Analyzer).
Device: Accu-Chek® Aviva Nano Meter/Accu-Chek® Aviva Test Strips — Study staff performed Blood Glucose (BG) tests with capillary fingerstick blood collected from subjects with diabetes. All meter BG results were compared with plasma results obtained with a reference laboratory glucose method (YSI Glucose Analyzer).
Device: Freestyle Lite® Meter and Test Strips with ZipwikTM tabs — Study staff performed Blood Glucose (BG) tests with capillary fingerstick blood collected from subjects with diabetes. All meter BG results were compared with plasma results obtained with a reference laboratory glucose method (YSI Glucose Analyzer).
Device: OneTouch® Ultra®2 / OneTouch® Ultra® Blue Test Strips — Study staff performed Blood Glucose (BG) tested with capillary fingerstick blood collected from subjects with diabetes. All meter BG results were compared with plasma results obtained with a reference laboratory glucose method (YSI Glucose Analyzer).
Device: One Touch® VerioTM Pro/One Touch® VerioTM Test Strips — Study staff performed Blood Glucose (BG) tests with capillary fingerstick blood collected from subjects with diabetes. All meter BG results were compared with plasma results obtained with a reference laboratory glucose method (YSI Glucose Analyzer).
Device: Truetrack® Meter/Truetrack® Test Strips — Study staff performed Blood Glucose (BG) tests with capillary fingerstick blood collected from subjects with diabetes. All meter BG results were compared with plasma results obtained with a reference laboratory glucose method (YSI Glucose Analyzer).

SUMMARY:
The purpose of this study was to test the performance of an investigational Bayer Blood Glucose (BG) meter and five additional Blood Glucose Monitoring Systems (BGMSs). The goal was to obtain glucose samples from subjects with diabetes across the meter operating ranges. A capillary sample was collected from each subject at 3 different times during the visit to obtain natural capillary blood samples with a range of glucose concentrations. Some blood samples were glycolyzed to lower the glucose concentration levels and glucose solution was added to other samples to raise glucose concentration levels. All meter BG results were compared with plasma results obtained with a reference laboratory glucose method (YSI Glucose Analyzer). All lancings and testing were performed by study staff.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of type 1 or type 2 diabetes mellitus
* 18 years of age or older
* Willing to follow all study procedures

Exclusion Criteria:

* Received an investigational drug or device within the last 30 days
* Current use or recent exposure to any prescription medication within 24 hours prior to screening that in the opinion of the investigator could have an influence on the subject's ability to participate in the study or on the performance on the test device
* Positive pregnancy test obtained at screening (test performed for females only, except if surgically sterile or three years past menopause)
* Hematocrit <32% or >55%
* Inadequate veins (in the opinion of the investigator or designated study staff) for venous blood withdrawal or intravenous catheter insertion
* Symptomatic coronary artery disease with a history of angina, or history of a myocardial infarction or coronary intervention (e.g. percutaneous transluminal coronary angioplasty [PTCA], stent placement) or coronary artery bypass graft (CABG) within the past 6 months
* Cerebrovascular accident within the past 6 months
* Diagnosis of the following diabetic autonomic neuropathies: symptomatic orthostatic hypotension, heart rate anomalies, gastroparesis
* Being treated for malignancy, except basal cell or squamous cell skin cancers
* Major surgical operation within 30 days prior to screening
* Active alcohol abuse or substance abuse (as judged by the principal investigator)
* Severe mental illness, mental incapacity, unwillingness or language barriers precluding adequate understanding or cooperation (as judged by principal investigator)
* Other medical conditions that would pose safety concerns, interfere with study conduct or seriously compromise study integrity, as judged by principal investigator (reason for exclusion will be clearly documented by investigator or designee)
* Working for a competitive medical device company, or having an immediate family member or someone who is not a family member but is living within the household of someone who works for such a company

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 146 (Actual)
Dates: Start 2012-05; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Leslie J Klaff, MD, Principal Investigator — Rainier Clinical Research Center Inc
Locations (1):
- Rainier Clinical Research Center Inc, Renton, Washington, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Intended BGM Users: Subjects were assigned to subgroups according to their initial glucose levels. SUBGROUP 1 goal:safely decrease subject glucose levels during the visit. SUBGROUP 2 goal: safely raise subject glucose levels. Also, blood samples were modified to obtain glucose concentrations across the needed glucose ranges while maintaining subject safety. Staff tested the blood samples using the 6 Blood Glucose Monitoring Systems. Bayer G3/Tatsu System;Accu-Chek® Aviva Nano Meter/Accu-Chek® Aviva Test Strips; Freestyle Lite® Meter and Test Strips with ZipwikTM tabs;OneTouch® Ultra®2 / OneTouch® Ultra® Blue Test Strips;One Touch® VerioTM Pro/One Touch® VerioTM Test Strips;Truetrack® Meter/Truetrack® Test Strips.
Period: Overall Study
Arm/Group | Intended BGM Users
Started | 146
Completed | 146
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Intended BGM Users
Number analyzed (Participants) | 146
Age, Continuous [Mean (Full Range); unit: years] | 53.0 [21 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 68
  Male | 78
Region of Enrollment [Number; unit: participants]
  United States | 146

OUTCOME MEASURES:

1. Primary Outcome: MAD Mean Absolute Value of the Difference Between Blood Glucose Meter (BGMS) Results and Corresponding YSI Blood Glucose (BG) Results in the Low BG Range(<70 mg/dL)
Description: Using samples with BG < 70 mg/dL, the Mean Absolute Value of the Differences Between BGM system readings and the YSI laboratory reference values were compared. MAD was calculated from the sum of all |(BG meter)-(BG reference)| assessments, divided by the number of assessments. Each evaluable sample was tested on all 6 BGMS, thus the same number of BG test results was analyzed for each BGMS intervention. Lower MAD value indicates smaller difference between meter value and the reference value. Higher MAD value indicates larger difference between meter value and the reference value.
Time Frame: 6 hours
Population: Same number (135) of BG results was possible for each BGMS. A capillary sample was collected from each subject at 3 different times during the visit to obtain natural capillary blood samples with a range of glucose concentrations. Subjects provided 85 unmodified capillary samples <70 mg/dL and 50 samples were modified by glycolyzing them.
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Units Other Than Participants: BG Results
Arm/Group | Intended BGM Users
Number analyzed (Participants) | 146
Number analyzed (BG Results) | 135
mg/dL
  Bayer G3/Tatsu System | 2.03 (0.430)
  Freestyle Lite® Meter | 2.77 (0.430)
  Accu-Chek® Aviva Nano Meter | 3.34 (0.419)
  One Touch® VerioTM Pro Meter | 4.53 (0.399)
  OneTouch® Ultra®2 Meter | 10.20 (0.416)
  Truetrack® Meter | 11.08 (0.416)

2. Secondary Outcome: MAD Mean Absolute Value of the Difference Between Blood Glucose Meter (BGMS) Results and Corresponding YSI Blood Glucose (BG) Results in the BG Range 70 to 180 mg/dL
Description: Using samples with BG 70 mg/dL to 180 mg/dL, the Mean Absolute Value of the Differences Between BGM system readings and the YSI laboratory reference values were compared. MAD was calculated from the sum of all|(BG meter)-(BG reference)| assessments, divided by the number of assessments. Each evaluable sample was tested on all 6 BGMS, thus the same number of BG test results was analyzed for each BGMS intervention. Lower MAD value indicates smaller difference between meter value and the reference value. Higher MAD value indicates larger difference between meter value and the reference value.
Time Frame: 6 hours
Population: Same number (172) of BG results was possible for each BGMS. A capillary sample was collected from each subject at 3 different times during the visit to obtain natural capillary blood samples with a range of glucose concentrations. Subjects provided all 172 capillary samples (70 to 180 mg/dL) and no samples were modified.
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Units Other Than Participants: BG results
Arm/Group | Intended BGM Users
Number analyzed (Participants) | 146
Number analyzed (BG results) | 172
mg/dL
  Bayer G3/Tatsu System | 4.29 (0.520)
  Accu-Chek® Aviva Nano Meter | 4.70 (0.527)
  One Touch® VerioTM Pro Meter | 5.18 (0.543)
  Truetrack® Meter | 9.71 (0.538)
  Freestyle Lite® Meter | 11.12 (0.532)
  OneTouch® Ultra®2 Meter | 11.13 (0.533)

3. Secondary Outcome: MAD Mean Absolute Value of the Difference Between Blood Glucose Meter (BGMS) Results and Corresponding YSI Blood Glucose (BG) Results in the BG Range >180 mg/dL
Description: Using samples with BG >180 mg/dL, the Mean Absolute Value of the Differences Between BGM system readings and the YSI laboratory reference values was compared. MAD was calculated from the sum of all |(BG meter)-(BG reference)| assessments, divided by the number of assessments. Each evaluable sample was tested on all 6 BGMS, thus the same number of BG test results was analyzed for each BGMS intervention. Lower MAD value indicates smaller difference between meter value and the reference value. Higher MAD value indicates larger difference between meter value and the reference value.
Time Frame: 6 hours
Population: Same number (231) of BG results was possible for each BGMS. A capillary sample was collected from each subject at 3 different times during the visit to obtain natural capillary blood samples with a range of glucose concentrations. Subjects provided 181 unmodified capillary samples >180 mg/dL and 50 samples were modified by adding glucose solution.
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Units Other Than Participants: BG Results
Groups:
- Intended BGM Users: Subjects were assigned to subgroups according to their initial glucose levels. SUBGROUP 1 goal: safely decrease subject glucose levels during the visit. SUBGROUP 2 goal: safely raise subject glucose levels. Also, blood samples were modified to obtain glucose concentrations across the needed glucose ranges while maintaining subject safety. Staff tested the blood samples using the 6 Blood Glucose Monitoring Systems.
Arm/Group | Intended BGM Users
Number analyzed (Participants) | 146
Number analyzed (BG Results) | 231
mg/dL
  Bayer G3/Tatsu System | 7.81 (1.137)
  Accu-Chek® Aviva Nano Meter | 8.77 (1.142)
  One Touch® VerioTM Pro Meter | 11.83 (1.143)
  OneTouch® Ultra®2 Meter | 18.78 (1.136)
  Truetrack® Meter | 26.47 (1.129)
  Freestyle Lite® Meter | 39.12 (1.116)

4. Secondary Outcome: Standard Deviations of BGMS Differences (Between BGM Meter Readings and the YSI Laboratory Reference Values Across the BG Range of All Evaluable Samples 21 mg/dL to 496 mg/dL)
Description: Variability of each meter system was determined by calculating the Standard Deviation derived from each meter's differences between Blood Glucose Meter (BGMS)results and corresponding YSI Blood Glucose (BG) results.
Time Frame: 6 hours
Population: Same numbers (538) of BG results were possible for each BGMS. A capillary sample was collected from each subject at 3 different times during the visit to obtain natural capillary blood samples with a range of glucose concentrations. Subjects provided 438 unmodified capillary samples and 100 samples were modified (21 to 496 mg/dL).
Measure: Number; unit: Standard Deviation
Units Other Than Participants: BG Results
Arm/Group | Intended BGM Users
Number analyzed (Participants) | 146
Number analyzed (BG Results) | 538
Standard Deviation
  One Touch® VerioTM Pro Meter | 7.02
  OneTouch® Ultra®2 Meter | 7.16
  Accu-Chek® Aviva Nano Meter | 7.57
  Bayer G3/Tatsu System | 8.05
  Truetrack® Meter | 9.88
  Freestyle Lite® Meter | 14.80

5. Secondary Outcome: Number of Subject Responses 'Strongly Agree' 'Agree' or 'Neutral' With Questionnaire Statements
Description: Subjects responded to statements about meter accuracy and diabetes management. Subject responses: 'Strongly Agree' 'Agree' 'Neutral' 'Disagree' or 'Strongly Disagree'or No Response. □1ACCURACY HELPS 1A-with my ability to talk with my HCP. 1B-my satisfaction with my self monitoring of diabetes. 1C-with my ability to manage my diabetes. 1D-prevent low BG. 1E-understand how food/exercise affects low BG. □2 I WOULD USE ONLY the meter and strips my insurance company pays for, even if a more accurate meter was available. □3 I USE MY CURRENT METER BECAUSE 3A-my HCP gave it to me. 3B-my insurance company covers the strips. 3C-I think it is the most accurate meter. □4 I WOULD SWITCH meters for a more accurate meter. □5BEING ABLE TO APPLY MORE BLOOD IS IMPORTANT 5A-as I have wasted test strips by not having enough blood to fill the strip 5B-as this would save test strips 5C-I would switch to a meter with this feature
Time Frame: 1 hour
Population: Since subjects had the option to provide No Response at all to a question, some questionnaire statements had less than 146 participant responses possible (see numbers in parentheses)
Measure: Number; unit: participants
Arm/Group | Intended BGM Users
Number analyzed (Participants) | 146
participants
  ACCURACY - QUESTION 1A (of 146) | 141
  ACCURACY - QUESTION 1B (of 146) | 136
  ACCURACY - QUESTION 1C (of 146) | 140
  ACCURACY - QUESTION 1D (of 145) | 138
  ACCURACY - QUESTION 1E (of 146) | 142
  QUESTION 2 (of 139) | 106
  QUESTION 3A (of 130) | 100
  QUESTION 3B (of 132) | 115
  QUESTION 3C (of 141) | 122
  QUESTION 4 (of 139) | 129
  QUESTION 5A (of 144) | 115
  QUESTION 5B (of 144) | 131
  QUESTION 5C (of 142) | 129

ADVERSE EVENTS:
Groups:
- Intended BGM Users: Subjects were assigned to subgroups according to their initial glucose levels. Subgroup 1 goal:safely decrease subject glucose levels during the visit. Subgroup 2 goal: safely raise subject glucose levels. Also, blood samples were modified to obtain glucose concentrations across the needed glucose ranges while maintaining subject safety. Staff tested the blood samples using the 6 Blood Glucose Monitoring Systems.
Arm/Group | Intended BGM Users
Serious Adverse Events (participants affected / at risk) | 0/146
Other Adverse Events (participants affected / at risk) | 5/146
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intended BGM Users (N=146)
Urinary tract infection (Renal and urinary disorders) | 1 (1) — Not study or device related, moderate severity
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Not study or device related,moderate severity
Upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 2 (2) — Not study or device related, mild
Nausea and vomiting (Gastrointestinal disorders) | 1 (1) — Not device related, moderate severity

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days